CLINICAL TRIAL: NCT05287009
Title: Optical Coherence Tomography Angiography (AngioVueTM, Optovue Inc., Fremont, Calif., USA) Changes in Patients With Epiretinal Membranes (ERM) With and Without Peeling of the Internal Limiting Membrane (ILM) - a Pilot Study
Brief Title: Optical Coherence Tomography Angiography (OCTA) Changes in Patients With Epiretinal Membranes (ERM) With and Without Peeling of the Internal Limiting Membrane (ILM)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 32-443 ex 19/20
Record Dates: First submitted 2022-03-10; First posted 2022-03-18 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Epiretinal Membrane of Both Eyes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ILM nonpeeling (Experimental)
  Interventions: Procedure: ILM nonpeeling
- ILM peeling (Other)
  Interventions: Procedure: ILM peeling

INTERVENTIONS:
Procedure: ILM nonpeeling — ILM is not peeled after ERM removal
  Arms: ILM nonpeeling
Procedure: ILM peeling — ILM is peeled after ERM removal
  Arms: ILM peeling

SUMMARY:
Main objective

The objective is to compare two surgical options in vitrectomies for epiretinal membranes using parameters of optical coherence tomography angiography.

Background

State of the art treatment for epiretinal membranes consists of pars plana vitrectomy, staining of the epiretinal membrane with a blue colouring dye and epiretinal membrane peeling. The vitrectomized space is filled with fluid (balanced salt solution) during the procedure and the fluid can optionally be replaced with air as a final step. After ERM peeling (but before the selection of the tamponade), the internal limiting membrane (the innermost layer of the retina) is either peeled as well or left untouched and the question which method should be preferred has been a hot topic in recent years. The investigators want to investigate possible effects of the used method (peeling vs. nonpeeling) on retinal perfusion parameters represented by OCTA. Two epiretinal membrane patient groups will therefore be formed: The first group's (group 1) ILM will be peeled, the second group's (group 2) ILM will not be peeled. After recruitement, patients will therefore be electronically randomized to one of the two groups. The groups will then be compared by the means of OCTA.

Study design

* Since there are no previous data on our research question, this investigation is defined as a pilot study.
* 40 patients with epiretinal membranes will be included. This appears to be a reasonable number given the incidence of epiretinal membranes. Previous studies that compared peeling versus nonpeeling in ERM used similar sample sizes. The detectable effect size was calculated at d = 0.91. We intend to complete this pilot study within 9 months.
* Randomization will be performed using electronic randomization. 20 patients each will be randomized to either group 1 or group 2.
* Both eyes in each patient will be imaged.
* No treatment decisions will be made based on OCTA findings. Treatment decisions will be made according to the clinic's standard of care.
* Three follow-up visits specific to the study are needed. These visits will be scheduled one week, one month and three months after surgery. All other preoperative and follow-up visits will be decided by the treating physician and follow the clinic standard of care.

Examinations

* Distance visual acuity using ETDRS (Early Treatment Diabetic Retinopathy Study) standard at 4 meters as per clinic standard of care.
* Tonometry as per clinic standard of care.
* Slit-lamp evaluation as per clinic standard of care.
* Arterial blood pressure.
* Axial eye length.
* Heidelberg Spectralis conventional OCT.
* The following 2 AngioVue scans will be taken:

A. One 3mm x 3mm, 304 x 304 A-scan OCTA of the macula B. One 6mm x 6mm, 304 x 304 A-scan OCTA of the macula

Hypothesis

The null hypothesis of our investigation indicates that there are no statistically significant differences in OCTA perfusion parameters based on the used option.

The alternative hypothesis states that there are statistically significant differences in OCTA perfusion parameters based on the used option.

Primary Objective

To demonstrate possible differences in OCTA perfusion parameters based on the used option.

Secondary Objectives

To assess the feasibility of the AngioVue optical coherence tomography angiography system in evaluating subtle changes in the retinal perfusion of patients with epiretinal membranes.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be able and willing to give informed consent.
* Patient must be over 18 and below 100 years of age.
* Patient must not have any significant media opacity which interferes with the examination.
* Patient must have an epiretinal membrane requiring surgery.

Exclusion Criteria:

* Unwilling or unable to provide informed consent
* Under 18 or over 100 years of age
* Significant media opacities
* Systemic pathologies making an examination difficult or cumbersome to the patient
* Secondary epiretinal membranes
* Bilateral epiretinal membranes
* Macular holes
* Lamellar holes
* Pseudo holes
* Glaucoma
* Diabetes
* Anisometropia > 2 diopters
* High myopia (spherical equivalent > 6 diopters and/or axial length > 26 mm
* Other retinal or ophthalmic pathologies except moderate cataract
* OCTA scan signal strength < 50
* Low image quality
* Failure of automatic layer segmentation

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2020-06-25 (Actual); Primary Completion 2022-03-09 (Actual); Study Completion 2022-03-09 (Actual)

PRIMARY OUTCOMES:
Superficial capillary plexus foveal avascular zone area | 3 months
  Superficial capillary plexus foveal avascular zone area (SCP FAZ) change (preoperative to postoperative). The SCP FAZ represents the area of the macula where blood vessels are not seen in OCTA under physiologic conditions. It has previously been reported that the FAZ narrows during ERM development and enlarges after ERM removal.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gabriel M, Djavid D, Innauer F, Ivastinovic D, Seidel G, Mayer-Xanthaki C, Ansari-Shahrezaei S, Wedrich A, Haas A. CHANGES OF OPTICAL COHERENCE TOMOGRAPHY ANGIOGRAPHY PARAMETERS AFTER INTERNAL LIMITING MEMBRANE PEELING COMPARED WITH NONPEELING IN EPIRETINAL MEMBRANE SURGERY. Retina. 2022 Oct 1;42(10):1867-1873. doi: 10.1097/IAE.0000000000003567. PMID 35976252